CLINICAL TRIAL: NCT05100277
Title: Impact of Oncotype DX® on Treatment Recommendation of for Early-stage Hormone Receptor-positive Breast Cancer and Its Economic Evaluation Under the Brazilian Society Perspective
Brief Title: Impact of Oncotype DX® on Treatment Recommendation and Its Economic Evaluation Under the Brazilian Society Perspective
Status: Completed | Type: Observational
Sponsor: Hospital Perola Byington (Other Government)
Collaborators: Fleury Laboratory (Unknown)
Responsible Party: Principal Investigator, Andre Mattar, PI, Hospital Perola Byington
Other Study IDs: 1/2020
Record Dates: First submitted 2021-05-18; First posted 2021-10-29 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer; Adjuvant Treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Costs and Cost Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Single arm: All patients will have the test
  Interventions: Genetic: Oncotype DX® Assay; Other: Cost

INTERVENTIONS:
Genetic: Oncotype DX® Assay — After surgery, tumoral tissue was used to perform Oncotype Dx®. Patients were evaluated and therapy recommendations - adjuvant chemotherapy (CT) plus hormone therapy (HT) or HT alone - were captured before and after revealing the test results. Results from TAILORx10 were used to guide decisions for or against CT for individual patients. Changes in treatment recommendations were obtained.
Other: Cost — Changes in treatment costs were estimated from Pérola Byington Hospital.

SUMMARY:
155 Pérola Byington Hospital patients presenting early stage luminal BC were submitted to Oncotype Dx® evaluation. Changes in treatment recommendations and costs were obtained from Pérola Byington Hospital. Oncotype DX® incorporation in the Brazilian Public Health System should be considered, as it results in high clinical impact for patient and high economic impact for health system, being a tool that safely and accurately delimits the subgroup of patients who really need AC.

DETAILED DESCRIPTION:
Background: It is known that there is significant over administration (and under administration) of adjuvant chemotherapy (AC) when standard clinical parameters (SCP) are used for patients diagnosed with early stage RE+ breast cancer (BC). Although absolute clinical benefit of AC may be modest, its toxicity and economic burden is highly significant; therefore, selecting appropriate patients for AC remains an important issue. Oncotype DX® identifies high-risk patients who are likely to benefit from AC, which otherwise might not be identified through SCP and low-risk patients who will not benefit from AC, thus avoiding toxicities and inherent risks. This study aimed to evaluate the impact of the Oncotype DX® test on treatment decisions in N0 and N1 early-stage breast cancer patients at a Public Brazilian hospital and to estimate the incremental cost-effectiveness ratio (ICER) and budget impact (BI) of incorporating Oncotype DX® under the perspective of the Brazilian Society.

Changes in treatment recommendations and costs will be obtained from Pérola Byington Hospital. Additional data will be obtained from literature. Medical costs (test, chemotherapy and adverse events), productivity loss, transportation and employment leave will be considered.

ELIGIBILITY:
Inclusion Criteria:

Women ≥ 18 years Early stage breast cancer, ER and/or PR positive with HER2 negative breast cancer.

Exclusion Criteria:

More than one operable primary breast tumor; Multifocal or multicentric tumors; 4 or more lymph node involvement; Metastatic breast cancer; Previous history of breast cancer; Invasive tumor <2 mm ; Performance status > 2 and / or other clinical factors that would make the patient a non-viable candidate for adjuvant chemotherapy; Previous hormonal or chemotherapy treatment; Current medical condition that would interfere with their ability to consent (psychiatric illness, for example)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with early stage breast cancer, positive ER and negative HER2 with negative lymph node or positive lymph node.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
The proportion of patients whose choice of treatment is changed as a result of Oncotype Test Low risk | up to 3 weeks
  Changes based on initial clinical measures
Economic evaluation | up to 5 years
  The costs of each scenario

CONTACTS AND LOCATIONS:
Locations (1):
- Andre Mattar, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All data will be available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available when the paper is published upon request
Access Criteria: described above